CLINICAL TRIAL: NCT04641195
Title: A Randomized Trial to Determine the Effect of Vitamin D and Zinc Supplementation for Improving Treatment Outcomes Among COVID-19 Patients in India
Brief Title: Vitamin D and Zinc Supplementation for Improving Treatment Outcomes Among COVID-19 Patients in India
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Foundation for Medical Research (Other); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Wafaie Fawzi, Professor of Nutrition, Epidemiology, and Global Health, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VR3- 172649
Record Dates: First submitted 2020-11-19; First posted 2020-11-23 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
Keywords: COVID-19; Vitamin-D3; Zinc; Nutrition support; Host-directed therapy; Clinical management; India
MeSH Terms: conditions — COVID-19 | interventions — Cholecalciferol; gluconic acid; Zinc; Vitamin D

STUDY DESIGN:
Intervention Model Description: The effect of both interventions (vitamin D or zinc) will be investigated simultaneously using a factorial design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo- Placebo (Placebo Comparator): Participants in the PLACEBO-PLACEBO group will receive a placebo vitamin D bolus at the hospital followed by placebo daily vitamin D maintenance doses and placebo daily zinc supplements.
  Interventions: Other: Placebo
- Vitamin D- Placebo (Experimental): Participants in the VITAMIN D-PLACEBO group will receive an actual vitamin D bolus at the hospital followed by actual daily vitamin D maintenance doses and daily placebo zinc supplements.
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)
- Placebo-Zinc (Experimental): Participants in the PLACEBO-ZINC group will receive a placebo vitamin D bolus at the hospital followed by placebo daily vitamin D maintenance doses and actual daily zinc supplements.
  Interventions: Dietary Supplement: Zinc (zinc gluconate)
- Vitamin D- Zinc (Experimental): Participants in the VITAMIN D-ZINC group will receive an actual vitamin D bolus at the hospital followed by actual daily vitamin D maintenance doses and actual daily zinc supplements.
  Interventions: Dietary Supplement: Zinc (zinc gluconate) & Vitamin D (cholecalciferol)

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (cholecalciferol) — 180,000 international units (IU) of vitamin D3 at enrollment, followed by 2000 IU once per day from enrollment to 8 weeks
  Arms: Vitamin D- Placebo
Dietary Supplement: Zinc (zinc gluconate) — 40mg of zinc gluconate taken once per day from enrollment to 8 weeks
  Arms: Placebo-Zinc
Dietary Supplement: Zinc (zinc gluconate) & Vitamin D (cholecalciferol) — 180,000 IU of vitamin D3 at enrollment, followed by 2000 IU of vitamin D3 and 40mg of zinc gluconate once per day from enrollment to 8 weeks
  Arms: Vitamin D- Zinc
Other: Placebo — Placebo vitamin D bolus at enrollment followed by placebo daily vitamin D maintenance doses and placebo daily zinc supplements.
  Arms: Placebo- Placebo

SUMMARY:
The purpose of this study is to assess the effect of vitamin D and/or zinc supplementation on improving COVID-19 treatment outcomes. The effects of vitamin D, zinc, and both vitamin D and zinc together will be investigated among COVID-19 patients in India.

DETAILED DESCRIPTION:
This study is a 2x2 factorial randomized double-blind, placebo-controlled trial to examine the effectiveness of vitamin D and zinc supplements as immune-based therapy among COVID-19 patients in India. The study is also examining the immunological response to COVID-19 and the effect of the intervention on specific biomarkers of immune and endothelial activation that are independent and quantitative predictors of severity and mortality in other severe infections. The primary aims are to determine the effect of vitamin D supplementation versus placebo on time to recovery among patients hospitalized with COVID-19; and to determine the effect of zinc supplementation versus placebo on time to recovery among patients hospitalized with COVID-19. As secondary aims, this study is also investigating the effect of vitamin D or zinc supplementation on all-cause mortality. necessity for assisted ventilation, individual symptoms duration, duration of hospital stay and biomarkers including vitamin D, Zinc, Interleukin 6 (IL-6), Angiopoietin-2, sTREM-1, immunoglobulin G (IgG) and immunoglobulin M (IgM).

Eligible individuals are randomly assigned to one of four groups: (1) Vitamin D (180,000 IU bolus at enrollment, followed by 2000 IU daily); (2) Zinc (placebo at enrollment followed by one daily dose of 40 mg); (3) Vitamin D and Zinc; or (4) Placebo. Daily supplements start at the hospital and continue after discharge for a total of 8 weeks. Active data collection occurs daily while patients are hospitalized and at least twice per week via telephone after discharge. A clinical exam occurs at 8 weeks and longer-term symptoms are assessed at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged >=18 years old
* Polymerase chain reaction (PCR) or Rapid Antigen Test (RAT)-confirmed infection with SARS-COV2
* Provide informed consent

Exclusion Criteria:

* Pregnancy
* Enrollment in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Time to recovery | Up to 8 weeks
  Defined as resolution of fever, cough and shortness of breath relative to baseline

SECONDARY OUTCOMES:
All-cause mortality | Up to 8 weeks
Necessity for assisted ventilation | Up to 8 weeks
Individual symptoms duration | Up to 8 weeks
Vitamin D | At 8 weeks
Zinc | At 8 weeks
Interleukin 6 (IL-6) | At 8 weeks
Angiopoietin-2 | At 8 weeks
sTREM-1 | At 8 weeks
Immunoglobulin M (IgM) | At 8 weeks
Immunoglobulin (IgG) | At 8 weeks
Duration of hospital stay | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Wafaie, MBBS, MPH, MS, DrPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (2):
- India (2):
  - Saifee Hospital, Mumbai, Maharashtra
  - King Edward Memorial (KEM) Hospital, Pune, Maharashtra

REFERENCES:
- [Derived] Partap U, Sharma KK, Marathe Y, Wang M, Shaikh S, D'Costa P, Gupta G, Bromage S, Hemler EC, Mistry N, Kain KC, Dholakia Y, Fawzi WW. Vitamin D and Zinc Supplementation to Improve Treatment Outcomes among COVID-19 Patients in India: Results from a Double-Blind Randomized Placebo-Controlled Trial. Curr Dev Nutr. 2023 Jul 11;7(8):101971. doi: 10.1016/j.cdnut.2023.101971. eCollection 2023 Aug. PMID 37560461
- [Derived] Martineau AR. Vitamin D in the prevention or treatment of COVID-19. Proc Nutr Soc. 2023 May;82(2):200-207. doi: 10.1017/S0029665122002798. Epub 2022 Nov 11. PMID 36366796
- [Derived] Sharma KK, Partap U, Mistry N, Marathe Y, Wang M, Shaikh S, D'Costa P, Gupta G, Bromage S, Hemler EC, Kain KC, Dholakia Y, Fawzi WW. Randomised trial to determine the effect of vitamin D and zinc supplementation for improving treatment outcomes among patients with COVID-19 in India: trial protocol. BMJ Open. 2022 Aug 29;12(8):e061301. doi: 10.1136/bmjopen-2022-061301. PMID 36038172